CLINICAL TRIAL: NCT03946345
Title: Iohexol for Measuring Renal Function
Acronym: HERO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL68547.091.18
Record Dates: First submitted 2019-05-03; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Acute Kidney Injury; Critically Ill Children
Keywords: Iohexol; Glomerular Filtration Rate
MeSH Terms: conditions — Acute Kidney Injury | interventions — Iohexol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * EDTA plasma samples
  * Urine samples
  * Whole blood samples (for future DNA-analysis)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Iohexol Inj 300 MG/ML — * Administration of iohexol: each 24 hours one bolus IV (1-5ml) during 72 hours
  * Blood samples are drawn for analysis of iohexol concentrations and other parameters of renal function at 2, 5 and 7 hours after administration
  * Urine is collected from catheter between 4 and 6 hours after adminstration to determine urine creatinine and iohexol concentrations
  Other Names: OMNIPAQUE 300

SUMMARY:
Approximately 25-35% of all children admitted to the paediatric intensive care unit (PICU) or neonatal intensive care unit (NICU) will develop Acute Kidney Injury (AKI) during the first seven days after admission. AKI is associated with a worse outcome, including an increased risk of mortality compared to patients without AKI. However, this AKI prevalence estimation is based on serum creatinine based glomerular filtration rate (eGFR), which is known to be inaccurate. The investigators postulate that measured GFR (mGFR) based on iohexol clearance in critically ill children will detect a higher prevalence of children with AKI than currently used methods based on endogenous markers. This study will additionally provide mechanistic knowledge on the relative contribution of GFR and renal transport to renal function in critically ill children.

DETAILED DESCRIPTION:
Primary objective: To determine the prevalence of AKI in critically ill children based on clearance of iohexol.

Secondary objectives:

1. To determine the prevalence of AKI in critically ill children using serum creatinine, creatinine clearance, cystatin C and/or blood urea nitrogen based eGFR equations as well as urinary iohexol clearances.
2. To determine serum Proenkephalin (PENK) levels in critically ill children.
3. To compare the prevalence of AKI when this diagnosis is based on plasma iohexol clearances with the prevalence of AKI based on serum creatinine, creatinine clearance, serum cystatin C, PENK and/or Blood Urea Nitrogen (BUN) based eGFR and to assess agreement between those methods
4. To determine risk factors for the development of AKI when based on iohexol clearance.

Exploratory endpoint: To explore the relationship of genetic variation with the development of AKI.

ELIGIBILITY:
Inclusion Criteria:

* 0-18 years of postnatal age
* >37 weeks of gestational age (for infants < one year postnatal age)
* Bodyweight >2500g
* Patients admitted to pediatric or neonatal intensive care unit
* PELOD-II (pediatric logistic organ dysfunction score, 2nd version) of 1 or higher (= at least one failing organ)
* Indwelling central line or arterial line in place for clinical purposes, or scheduled regular blood work for clinical reasons (at least once a day)
* Informed written consent

Exclusion Criteria:

* Known medical history of allergic reaction to injection of iodinated contrast material
* Receiving renal replacement therapy
* Language or cognitive inability of parents/caregivers to understand written and oral informed consent.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 105 critically ill children admitted to the pediatric intensive care unit or neonatal intensive care unit from the Radboudumc with at least one failing organ.
Sampling Method: Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of AKI in critically ill children based on iohexol plasma clearance | 72 hours
  AKI will be defined by using age-specific reference values of GFR. Based on their standard deviations (SD), three groups are defined:
  * Stage 1: mean -1 SD > GFR < mean -1.5 SD
  * Stage 2: mean -1.5 SD> GFR < mean -2 SD
  * Stage 3: GFR < mean -2 SD
  Patients will be grouped according whether they lack AKI or have AKI (either stage 1, 2 or 3). When a patient will be classified as having AKI at one moment and not fulfilling the AKI-criteria at another, or classified into different stages of AKI within one day, the highest stage of the 72 hours will be used for analysis.

SECONDARY OUTCOMES:
Prevalence of AKI using serum creatinine, creatinine clearance, urinary iohexol, serum cystatin C, serum PENK and/or blood urea nitrogen based eGFR equations. | 72 hours
  Classification of AKI based on serum creatinine levels:
  * Stage 1: serum creatinine concentration >150% of median age specific reference value.
  * Stage 2: serum creatinine concentration >200% of median age specific reference value.
  * Stage 3: serum creatinine concentration >300% of median age specific reference value.
  Creatinine clearance: CrCl(ml/min/1.73m2) = (urine volume × urine creatinine × 1.73)/ (serum creatinine × 120 minutes × body surface area)
  AKI classification based on serum cystatin C levels will be similar to classification based on serum creatinine levels
  Urinary iohexol clearance: Ku(X)(t)=dXu/dt & Cl(u)=dXudt/AUCpdt
  AKI will be classified based on eGFR calculated by the CKiD Schwartz Equation
  Data will be analysed for the overall 72 hour period, using the highest grade of AKI during the study duration, as well as per 24 hour period.
Serum PENK levels, in relation to iohexol based GFR-measurements in critically ill children. | 72 hours
Agreement between diagnosis of AKI when based on iohexol clearance compared to diagnosis based on serum creatinine levels | 72 hours
Agreement between diagnosis of AKI when based on iohexol clearance compared to diagnosis based on creatinine clearance | 72 hours
Agreement between diagnosis of AKI when based on iohexol clearance compared to diagnosis based on serum cystatin C levels | 72 hours
Agreement between diagnosis of AKI when based on iohexol clearance compared to diagnosis based on serum PENK levels | 72 hours
Agreement between diagnosis of AKI when based on iohexol clearance compared to diagnosis based on CKiD Schwartz Equation (Serum Creatinine, BUN and Cytatin C) | 72 hours
Risk factors for the development of AKI when based on iohexol clearance. | 72 hours

OTHER OUTCOMES:
To explore the relationship of genetic variation with the development of AKI. | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Saskia N De Wildt, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No